CLINICAL TRIAL: NCT00435617
Title: Clinical Assessment of a Massed Practice Therapy Device
Brief Title: Study of Hand Therapy 3 to 24 Months After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinetic Muscles (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Koeneman, Chief Science Officer, Kinetic Muscles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44HD041805 (NIH); R44HD041805 (NIH)
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Cerebrovascular Accident
Keywords: stroke rehabilitation; stroke therapy; hand therapy; stroke; cerebrovascular stroke; cerebral stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Hand Mentor
  Interventions: Device: Hand Mentor

INTERVENTIONS:
Device: Hand Mentor — Use of the Hand Mentor therapy device at home for 6 weeks. Therapy programs include spasticity reduction, motor control, and emg biofeedback for encouraging activity.
  Other Names: Hand Mentor Home

SUMMARY:
The primary aim of this study is to investigate the effectiveness of the use of a robotic hand therapy device in the home environment. We hypothesize that the therapy group will improve hand function more than a customary and usual care group.

DETAILED DESCRIPTION:
Many stroke survivors have significant limitations of upper extremity function which impacts many important activities such as eating, dressing and personal care. Studies show that to be effective in increasing functional independence, therapy must involve active participation of the patient and repetitive training. Robotic therapy offers a means of transferring some of this essential, but time consuming, therapy into the home. Seventy subjects (3 to 12 months post stroke)are being randomized to a control group that utilizes an innovative robotic hand therapy device in the home for three months or a control group that receives no device treatment. Clinical motor function and quality of life measures will compare the groups before intervention, immediately after, and 3 months later. The control group will receive device treatment for 3 months following their final evaluation. The results will provide valuable data on the ability of monitored home therapy to provide effective treatment. This project has the potential to increase the availability of effective rehabilitation techniques to patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 24 months post stroke
* Able to extend wrist and fingers at least 10 degrees
* Functional hearing and vision
* Able to follow instructions
* Lives at home, not institution
* Stable medications for 3 months

Exclusion Criteria:

* Excessive cognitive impairments
* Taking/Receiving medicines/shots to make arm/hand less stiff
* Severe pain in the impaired arm
* Stroke was more than 24 months ago

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Initial, 6 wks, 12 wks, 16 wks, 52 wks

SECONDARY OUTCOMES:
Compliance with recommended use | 6 wks, 12 wks
Fugl-Meyer Test | Initial, 6 wks, 12 wks, 16 wks, 52 wks
Stoke Impact Scale | Initial, 6 wks, 12 wks, 16 wks, 52 wks

CONTACTS AND LOCATIONS:
Overall Officials: James B Koeneman, Ph.D., Principal Investigator — Kinetic Muscles, Inc.; Steven L Wolf, Ph.D., PT, Study Director — Emory University Medical School; Richard Herman, MD, Study Director — Banner Good Samaritan Medical Center
Locations (2):
- United States (2):
  - Arizona State University, College of Nursing & Healthcare Innovation, Phoenix, Arizona
  - Emory University, Atlanta, Georgia

REFERENCES:
- [Background] Frick EM, Alberts JL. Combined use of repetitive task practice and an assistive robotic device in a patient with subacute stroke. Phys Ther. 2006 Oct;86(10):1378-86. doi: 10.2522/ptj.20050149. PMID 17012642